CLINICAL TRIAL: NCT05501041
Title: Quantification of Symptom Relief Following Percutaneous Ablation of the Thyroid
Brief Title: Measuring Symptom Relief After Radiofrequency Ablation of the Thyroid
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas D. Atwell, Principal Investigator, Mayo Clinic
Other Study IDs: 22-007581
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Thyroid
Keywords: Thyroid Radiofrequency Ablation Procedure
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to measure the impact of thyroid radiofrequency ablation procedure on patients with thyroid-related symptoms using a modified pre-existing scoring system.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing Radiofrequency Ablation (RFA) for symptomatic thyroid nodule(s).

Exclusion Criteria:

- Decline to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing ablation for symptomatic thyroid nodule(s)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms before and after ablation | Baseline and 1-, 3-, 6-, 12-, 18-, and 24-months following treatment
  Measured using a modified 6-item SYS questionnaire that objectively measures patient symptoms on a scale of 0=none, 1=moderate, 2=severe

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Atwell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials